CLINICAL TRIAL: NCT02104453
Title: Comparative Evaluation of One-handed E-C Clamp Mask Holding Technique, Two-handed Mask Ventilation With Jaw Thrust, and Two-handed Mask Ventilation With Triple Airway Maneuver in the Unconscious Apneic Person
Brief Title: Comparative Evaluation of Three Airway Maneuvers in the Unconscious Apneic Person
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hung Chan, Anesthesiology Department, Tri-Service General Hospital, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-103-05-029; WChan (Registry Identifier: WChan)
Record Dates: First submitted 2014-03-28; First posted 2014-04-04 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Airway Morbidity
Keywords: airway maneuver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- E-C clamp mask holding technique (Experimental): the airway maneuver that press the mask against the patient's face (using the "C" of our thumb and forefinger) while pulling the jaw forward (using the "E" of our other fingers behind the mandible), and leaves one hand free to squeeze the bag.
  Interventions: Procedure: airway maneuver
- two-handed ventilation with jaw thrust (Experimental): the airway maneuver performed with thumbs point toward feet, palms press down and other fingers perform jaw thrust
  Interventions: Procedure: airway maneuver
- triple airway maneuver (Experimental): the airway maneuver performed with two-handed mask ventilation, jaw thrust and head-tilt chin-lift technique
  Interventions: Procedure: airway maneuver

INTERVENTIONS:
Procedure: airway maneuver — Three-period crossover study: During general anesthesia induction, subjects are assigned to one of the 6 airway maneuver sequences (ABC, CAB, BCA, ACB, CBA, or BAC) in accordance with a randomization schedule. Each maneuver is performed 5 times in a period.
  Airway maneuver A: E-C clamp mask holding technique; Airway maneuver B: two-handed mask ventilation with jaw thrust airway maneuver; Airway maneuver C: two-handed mask ventilation with triple airway maneuver(combine jaw thrust and head tilt chin lift)

SUMMARY:
One-handed E-C clamp mask holding technique, two-handed mask ventilation with jaw thrust, and two-handed mask ventilation with triple airway maneuver are three common airway management maneuvers. Sniffing position may improve ventilation between these three maneuvers. The investigators hypothesize that ventilation efficiency may be different between these three maneuvers whether the patient is in sniffing position or neutral position. The investigators would like to quantify this effect by measuring the expired tidal volume, airway pressure, EtCO2 slope and hemodynamic change between these three maneuvers during anesthesia induction.

DETAILED DESCRIPTION:
Mask ventilation is considered a important skill for airway management during general anesthesia induction and for apneic unconscious patients. One-handed E-C clamp mask holding technique, two-handed mask ventilation with jaw thrust, and two-handed mask ventilation with triple airway maneuver are three common airway management maneuvers. However, the efficiency of ventilation between these three maneuvers has to be clarified. Besides, whether sniffing position or neutral position may improve ventilation between these three maneuvers is to be determined. The investigators will collect airway parameters of the patients receiving general anesthesia and measure the expired tidal volume, airway pressure, EtCO2 slope and hemodynamic change between these three maneuvers during anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* adult patients(ASA I-III) scheduled for elective surgery requiring general anesthesia with endotracheal intubation.

Exclusion Criteria:

* pneumothorax
* SpO2<96%(without additional oxygen supply)
* vocal cord palsy
* congenital airway abnormality
* facial trauma or deformity
* acute upper airway disease
* inadequate fasting time
* neck or potential cervical spine disease
* temporal-mandible joint abnormality
* head and neck tumor
* status post radiotherapy
* pregnancy
* long term sedative or opioid drug use
* patient refuse

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Air exchange | during anesthesia induction
  Expired tidal volume, end tidal CO2 slope, peak inspiratory pressure between one-handed E-C clamp mask holding technique, two-handed mask ventilation with jaw thrust, and two-handed mask ventilation with triple airway maneuver

SECONDARY OUTCOMES:
Hemodynamic change | during anesthesia induction
  blood pressure and heart rate variability during ventilation between one-handed E-C clamp mask holding technique, two-handed mask ventilation with jaw thrust, and two-handed mask ventilation with triple airway maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Chan, doctorate, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan